CLINICAL TRIAL: NCT02375581
Title: A Phase II Study of Icotinib With Concurrent Radiotherapy in Elderly Patients With Esophageal Cancer
Brief Title: Phase II Study of Icotinib With Concurrent Radiotherapy in Elderly Patients With Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HZFH CA15-01
Record Dates: First submitted 2015-02-16; First posted 2015-03-02 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Esophageal Cancer
Keywords: Radiotherapy; Icotinib
MeSH Terms: conditions — Esophageal Neoplasms | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Icotinib & Radiotherapy (Experimental): Icotinib, 125mg, Po, Tid, during the course of radiotherapy; Thoracic radiotherapy, 50-60Gy, conventional fraction, 3D-CRT/IMRT.
  Interventions: Drug: Icotinib; Radiation: Thoracic radiotherapy
- Radiotherapy alone (Active Comparator): Thoracic radiotherapy alone, 50-60Gy, conventional fraction, 3D-CRT/IMRT.
  Interventions: Radiation: Thoracic radiotherapy

INTERVENTIONS:
Drug: Icotinib — 125mg, Po, TID during RT
  Other Names: Conmana
  Arms: Icotinib & Radiotherapy
Radiation: Thoracic radiotherapy — involved-Field irradiaton without elective nodal irradiation

SUMMARY:
To investigate the efficacy and toxicity of EGFR tyrosine-kinase inhibitor (Icotinib) with concurrent radiotherapy in older patients with esophageal cancer.

DETAILED DESCRIPTION:
Older patients with esophageal cancer have been correlated with poor prognosis because of having little chance to receive aggressive local therapy, including surgery or concurrent chemoradiotherapy. EGFR is overexposed in most of the cases. In this phase II trial, the efficacy and toxicity of EGFR tyrosine-kinase inhibitor (Icotinib) with concurrent radiotherapy will be investigated in this setting.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed esophageal carcinoma
2. Stage I～Iva By EUS and CT/MRI, without contraindication for radical radiotherapy
3. Aged ≥ 70 and < 85 years, behavioral status evaluation ECOG scores 0-2
4. In 7 days after being screened, subjects should follow the status: WBC ≥ 3.0 x 10^9/L; ANC ≥ 1.5x 10^9/L; PLT ≥ 80 x 10^9/L; Hb ≥ 90 g/L; serum Cr ≤ ULN; serum bilirubin ≤ 1.5 ULN; ALT/AST ≤ 1.5 ULN
5. Subjects should sign for the informed consent
6. Subjects should perform good compliance

Exclusion Criteria:

1. Patients who have or are currently undergoing additional chemotherapy, radiation therapy or targeted therapy
2. Complete obstruction of the esophagus, or patients who have the potential to develop perforation
3. Patients with a history of malignancy (except that skin carcinomas or in situ breast cancer, oral cancer and cervical cancer with expected survival ≥2 years
4. Patients who have multiple foci esophageal carcinomas
5. Patients who are/were given any other medicine tests currently/in last 4 weeks
6. Experienced hypersensitiveness with similar medicine or other kinds of bio-medicines
7. Patients who have complications as following:

(1) Uncontrolled angina and heart failure, have a history of hospitalization in 3 months; (2) A history of myocardial infarction in the past 6 months; (3) There is a need for antibiotic treatment of acute bacterial or fungal infection; (4) Chronic obstructive pulmonary disease, or other lung disease requiring hospitalization; (5) Drug addiction, alcoholism and AIDS disease or long-term virus carriers; (6) Uncontrollable seizures, or loss of insight because of mental illness.

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | 2 years

SECONDARY OUTCOMES:
incidence rates of radiation-related pneumonitis and esophagitis | within the 3 months after the initiation of RT

CONTACTS AND LOCATIONS:
Overall Officials: Shixiu Wu, MD, Principal Investigator — Hangzhou Cancer Hospital
Locations (1):
- Hangzhou Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Luo H, Jiang W, Ma L, Chen P, Fang M, Ding L, Hua Y, Du D, Jing Z, Xie R, Song Y, Wang J, Zhou R, Tian Z, Wu S. Icotinib With Concurrent Radiotherapy vs Radiotherapy Alone in Older Adults With Unresectable Esophageal Squamous Cell Carcinoma: A Phase II Randomized Clinical Trial. JAMA Netw Open. 2020 Oct 1;3(10):e2019440. doi: 10.1001/jamanetworkopen.2020.19440. PMID 33026449